CLINICAL TRIAL: NCT01440543
Title: Combination of Water Immersion and Carbon Dioxide Insufflation for Minimal Sedation Colonoscopy - a Prospective, Randomized, Single-center Trial
Brief Title: Combination of Water Immersion and Carbon Dioxide Insufflation for Minimal Sedation Colonoscopy
Acronym: Water/CO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitkovice Hospital (Other)
Responsible Party: Principal Investigator, Premysl Falt MD, Principal Investigator, Vitkovice Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DDC VN 01
Record Dates: First submitted 2011-09-19; First posted 2011-09-26 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2012-12

CONDITIONS: Colonoscopy
Keywords: colonoscopy; water immersion; CO2 insufflation; patients referred for diagnostic outpatient colonoscopy; (screening, surveillance, symptoms); patient discomfort associated with diagnostic colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Water/CO2 (Experimental): water immersion during colonoscope insertion and CO2 insufflation during colonoscope withdrawal
  Interventions: Procedure: Water immersion insertion AND CO2 insufflation
- Water/Air (Experimental): Water immersion during colonoscope insertion and air insufflation during colonoscope withdrawal
  Interventions: Procedure: Water immersion insertion
- CO2/CO2 (Experimental): CO2 insufflation during both colonoscope insertion and withdrawal
  Interventions: Procedure: CO2 insufflation
- Air/Air (No Intervention): room air insufflation during both colonoscope insertion and withdrawal

INTERVENTIONS:
Procedure: Water immersion insertion AND CO2 insufflation — * room temperature water infused by water pump into the colon just to facilitate scope insertion
  * CO2 insufflation by CO2 insufflation system during colonoscope withdrawal and mucosal inspection
  Arms: Water/CO2
Procedure: Water immersion insertion — * room temperature water infused by water pump into the colon just to facilitate scope insertion
  * standard room air insufflation during colonoscope withdrawal and mucosal inspection
  Arms: Water/Air
Procedure: CO2 insufflation — - CO2 insufflation by CO2 insufflation system during both colonoscope insertion and withdrawal
  Arms: CO2/CO2

SUMMARY:
Water immersion insertion and carbon dioxide (CO2)instead of room air insufflation as alternative colonoscopy techniques have been documented to decrease patient discomfort during and after the procedure.

This prospective, randomized, single-center trial was designed to evaluate whether the combination of water immersion during insertion and CO2 insufflation during withdrawal (Water/CO2)for minimal sedation colonoscopy (2 mg of midazolam i.v.)is superior to the other colonoscopy methods (Water/Air, CO2/CO2, Air/Air).

ELIGIBILITY:
Inclusion Criteria:

* men and women older than 18 years referred for diagnostic outpatient colonoscopy
* provided written consent

Exclusion Criteria:

* history of colorectal surgery
* known diagnosis of inflammatory bowel disease
* chronic benzodiazepine use
* refusal of minimal sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Premysl Falt, MD, Principal Investigator — Digestive Diseases Center, Vitkovice Hospital, Ostrava, Czech Republic
Locations (1):
- Digestive Diseases Center - Vitkovice Hospital, Ostrava, Czechia

REFERENCES:
- [Result] Falt P, Liberda M, Smajstrla V, Kliment M, Bartkova A, Tvrdik J, Fojtik P, Urban O. Combination of water immersion and carbon dioxide insufflation for minimal sedation colonoscopy: a prospective, randomized, single-center trial. Eur J Gastroenterol Hepatol. 2012 Aug;24(8):971-7. doi: 10.1097/MEG.0b013e3283543f16. PMID 22569079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * recruitment process between January and June 2011
  * outpatients referred to our endoscopy unit for diagnostic colonoscopy
Pre-assignment Details: * a total of 548 patients were assessed for eligibility
  * a total of 420 patients were randomized after exclusion of 128 subjects because of not fulfilled inclusion criteria
  * a total of 404 patients were analyzed after exclusion of 16 subjects (poor bowel preparation, IBD, argon plasmacoagulation, endoscopic resection or malignant obstruction)
Period: Overall Study
Arm/Group | Water/Air | CO2/CO2 | Water/CO2 | Air/Air
Started | 106 | 105 | 102 | 107
Completed | 102 | 101 | 100 | 101
Not Completed | 4 | 4 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Water/Air | CO2/CO2 | Water/CO2 | Air/Air | Total
Number analyzed (Participants) | 106 | 105 | 102 | 107 | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 55 | 60 | 54 | 58 | 227
  >=65 years | 51 | 45 | 48 | 49 | 193
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (13.9) | 59.4 (14.5) | 58.2 (13.4) | 58.7 (13.8) | 59.2 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 52 | 49 | 51 | 202
  Male | 56 | 53 | 53 | 56 | 218
Region of Enrollment [Number; unit: participants]
  Czech Republic | 106 | 105 | 102 | 107 | 420

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Minimal Sedation Colonoscopy
Description: Successful minimal sedation colonoscopy using assigned technique was defined as reaching the caecum without switch to another insertion method and / or without additional sedation beyond the initial administration of 2 mg of midazolam.
Time Frame: six months
Reporting Status: Not Posted

2. Secondary Outcome: Patient Comfort During the Procedure and During First 24 Hours After Procedure
Description: Comfort was assessed using a 18-point questionnaire form based on 0-6 continuous scale (0 = best, 6 = worst)- abdominal pain during, 30 minutes, 3, 12 and 24 hours after the procedure, bloating duringm 30 minutes, 3, 12 and 24 hours after the procedure, flatus during, 30 minutes, 3, 12 and 24 hours after the procedure, impact on patient´s daily activities during first 24 hours after the procedure, willingnes to repeat the colonoscopy and overall satisfaction with the procedure
Time Frame: six months
Reporting Status: Not Posted

3. Primary Outcome: Success Rate of Minimal Sedation Colonoscopy
Description: A succesful colonoscopy using assigned technique was defined as reaching the caecum without switching to another insertion method and without additional sedation beyond the initial 2 mg of midazolam. Any time the further insertion of the scope was not possible, the patient reported pain level > 3 using a 7-point Likert scale [7] (0 = no pain, 6 = intolerable pain) or demanded additional sedation, the endoscopist preferentially switched to the other insertion technique. Enhanced sedation was used in case the other technique had not been successful.
Time Frame: 6 months
Population: Statistical power was calculated for the primary endpoint. A sample size of 145 subjects per insertion arm was calculated using two-tailed α = 0,05, β = 0,05, assuming that 80% versus 60% success rate in the water (Water/CO2 and Water/Air) and gas (CO2/CO2 and Air/Air) insertion arms would have been clinically relevant.
Measure: Number; unit: percentage of all participants
Arm/Group | CO2/CO2 | Water/Air | Water/CO2 | Air/Air
Number analyzed (Participants) | 102 | 100 | 101 | 101
percentage of all participants | 82.4 | 97 | 97 | 84.2

ADVERSE EVENTS:
Arm/Group | Water/Air | CO2/CO2 | Water/CO2 | Air/Air
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
There were no procedure- or sedation-related complications recorded in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No